CLINICAL TRIAL: NCT05091814
Title: : Post-operative Prevalence of Trismus in Patients With Maxillary Cancer With and Without Radiation Therapy in the Egyptian Population.(a Cross Sectional Study)
Brief Title: Prevalence of Trismus in Patients With Maxillary Cancer With and Without Radiation Therapy in the Egyptian Population.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Mohamed Diaa Eldin Erfan, : Post-operative Prevalence of trismus in patients with maxillary cancer with and without radiation therapy in the Egyptian population.(a cross sectional study), Cairo University
Other Study IDs: 10621
Record Dates: First submitted 2021-09-26; First posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: Maxillary Neoplasms
Keywords: surgery , Trismus, Oral
MeSH Terms: conditions — Maxillary Neoplasms; Trismus | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Radiotherapy (Yes or no) - Exercise (YES or NO): with or without radiotherapy
  Interventions: Radiation: radiotherapy
- MMO (in mm): with or without radiotherapy

INTERVENTIONS:
Radiation: radiotherapy — patients who recieved radiotherapy after surgical removal of the tumor
  Groups: Radiotherapy (Yes or no) - Exercise (YES or NO)

SUMMARY:
This study aims at evaluating the prevalence of trismus among maxillary cancer patients in the Egyptian population and the effect of radiotherapy on the occurrence of trismus.

DETAILED DESCRIPTION:
The enrolled participants who meet the eligibility criteria and signed the informed consent of participation in the study will undergo clinical examination to determine the maximum mouth opening after performing surgery only and /or after radiotherapy in case of adjuvant therapy

the maximum mouth opening will be measured in (mm) by using a digital caliper device and will be recorded in the patient sheet,

reading of less than 35mm will be considered trismus while above 35mm or more will be considered normal (NO trismus)

ELIGIBILITY:
Inclusion Criteria:

* patients with maxillary cancer

Exclusion Criteria:

* patients under 18 yrs .
* patients with TMJ disorders before surgery
* patients on chemotherapy
* - Tumors in other sites( Tongue , buccal mucosa , salivary glands, mandible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with maxillary cancer attending faculty of dentistry ,CU and the national cancer institute.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2021-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
% prevalence | 1 year
  Trismus prevalence in percent

SECONDARY OUTCOMES:
MMO | 1 year
  maximum mouth opening

CONTACTS AND LOCATIONS:
Overall Officials: Gamal Ashour, Study Director — National Cancer Institute (NCI)
Locations (1):
- Cairo University, Cairo, Haram, Egypt

IPD SHARING:
Plan to Share IPD: Yes
the results of the study will be available at the college library for the researchers to benefit from.
Supporting Information: CSR
Time Frame: 1-2 years
Access Criteria: Free access
URL: http://clinicaltrials.gov

REFERENCES:
- [Result] van der Geer SJ, van Rijn PV, Kamstra JI, Langendijk JA, van der Laan BFAM, Roodenburg JLN, Dijkstra PU. Prevalence and prediction of trismus in patients with head and neck cancer: A cross-sectional study. Head Neck. 2019 Jan;41(1):64-71. doi: 10.1002/hed.25369. Epub 2018 Dec 18. PMID 30561067